CLINICAL TRIAL: NCT04171648
Title: Effect of Dry Roasted Peanuts and Boiled Peanuts on Glycemic Control
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 Pandemic halted my study due to exposure risks.
Sponsor: North Carolina State University (Other)
Responsible Party: Principal Investigator, Brooke Wilson, Master of Science Nutrition (Thesis) Graduate Student, North Carolina State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 19049
Record Dates: First submitted 2019-11-15; First posted 2019-11-21 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus; Glycemic Control
Keywords: diet management; weight management
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Half the subjects will receive the roasted peanut treatment and the other half will receive the boiled peanut treatment for two weeks, then both will have a week wash out, and then each group will switch to the opposite treatment for two weeks.
Masking Description: The nature of the participants eating (whole food) peanut samples roasted or boiled allows no way for the participants or the investigators to be masked from the two interventions. The care provider does not apply in this study and the outcomes assessor will be the same individual as the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roasted Peanut Group 1 (Experimental): Arm 1 is the arm of participants that will receive the roasted peanut treatment first and then will crossover to the boiled peanut treatment.
  Interventions: Other: Roasted Peanut Treatment; Other: Boiled Peanut Treatment
- Boiled Peanut Group 1 (Experimental): Arm 2 is the arm of participants that will receive the boiled peanut treatment first then will crossover to the roasted peanut treatment.
  Interventions: Other: Roasted Peanut Treatment; Other: Boiled Peanut Treatment

INTERVENTIONS:
Other: Roasted Peanut Treatment — The subjects will consume 2 ounces or ~48 grams of roasted in shell peanuts a day for two weeks.
Other: Boiled Peanut Treatment — The subjects will consume 2 ounces or ~48 grams of boiled peanuts a day for two weeks.

SUMMARY:
Research on glycemic control related to nuts or whole snack foods has focused primarily on tree nuts. Different processing and cooking methods have not been comprehensively analyzed to observe the effect on nutrient quality, bioavailability, or digestive absorption in peanuts. There is little to no research surrounding the nutrition of boiled peanuts so it may be of interest to compare boiled to roasted peanuts in terms of glycemic control. Peanuts have been shown to have a similar beneficial effect on glycemic control while being more financially accessible than almonds. Glycemic control could be improved based on the low glycemic index, high fiber, lipid, and or protein content of peanuts. The acute trial (phase 1) will investigate the impact of preprandial peanut consumption on glycemic response. The participants will complete an oral glucose tolerance test for both roasted and boiled peanuts. The long term study (phase 2&3) consists of participants consuming one serving per day of boiled or roasted peanuts in a four week crossover trial to observe any long term impact of daily peanut snacking on glycemic control. (Wash out weeks occurring between all trials.) At the conclusion of phase 2 & 3 an oral glucose tolerance test will be executed. The subjects will self record a exercise/step count and diet dairy, weight and waist to hip ratio will be measured weekly. The study will aim for a male and/or female healthy population from 18-65 years of age at NCSU.

DETAILED DESCRIPTION:
Participants will be recruited via flyers, oral presentations, and emails. The recruitment methods will briefly describe the study, eligibility, and compensation asking potential subjects to contact Brooke Wilson for more information (by email) in which Brooke will respond by email with the time and place of the informational meeting that will include the screening process of the health screening questionnaire. The questionnaire will be attached/included in the response email so the interested individual may see if they are eligible before coming to the meeting. The health screen questionnaire will not be kept by the research team, if the participant says "yes" to any question they are determined to be not eligible and investigators will shred all health questionnaires and no participant needs to write their name on a questionnaire. At the informational meeting the study protocol, schedule of phases including total hours required, risks and benefits, and compensation will be discussed as well as physical copy of the consent form will be given to review. A health screening questionnaire will be provided and the subject will fill it out privately and/or ask questions if required. Those individuals who meet the initial eligibility criteria included in the questionnaire and voluntarily signs the consent form will be asked to schedule an oral glucose tolerance test as a following separate meeting that will determine if their glycemic response meets the final eligibility. Oral Glucose Tolerance Test ELIGIBILITY: (1 morning duration ~3 hours in lab) The investigators will inform participants at the meeting (also described in consent form) that the test will start early in the morning when they have not eaten anything since the previous evening, or at least 6 to 8 hours in this fasted state. The screening will measure fasting blood glucose (one reading of blood glucose before the test begins) and a glucose tolerance test will be done to rule out subjects with insulin resistance. A glucose tolerance test measures changes in blood glucose over a 2-hr period after consuming a glucose drink containing 50 g of glucose. Blood samples will be taken at 10, 20, 30, 40, 50, 60, 75, 90, 105, and 120 min after consuming the treatments using a glucometer to take capillary blood samples (finger-pricks); (The "oral" descriptor of the test refers to the fact that the individual orally ingests a 50 gram glucose drink which mimics a standard meals spike in the blood glucose response. The "oral" differentiates the method of administering glucose, such as in other cases the glucose can be injected intravenously instead of ingested through food or drink form. All glucose tolerance tests will monitor blood glucose by using continuous glucometers or drawing blood in increments of time.) No participant will be left alone during the oral glucose tolerance test, during all tests Brooke Wilson and a second research team member will be with the participants. Brooke Wilson and staff will measure height, hip to waist ratio and weight of the subjects. These measurements will be taken in a private room, with two staff at all time that are the same gender as the participant, and everyone will be fully clothed during all times. Professors will not take any measurements. Height and weight are measured to calculate body mass index over the course of the study to observe any weight changes that may be associated with a change in diet. Measuring hip to waist ratio will give a more accurate idea of weight distribution, general health, and risk of certain diseases. Subjects with glucose responses considered normal/healthy will be invited to continue in the study. It is possible that a participant could pass the health screen questionnaire, sign the consent form, and then fail the oral glucose tolerance test in which they will not be allowed to continue in the study and will not be compensated in any form. The consent form must be signed before the oral glucose tolerance test to determine eligibility for the participants safety and awareness of risks. The oral glucose tolerance test conducted for eligibility will also function as a baseline reading for those participants who complete the study. The health screening questionnaire will be shredded immediately after the subjects agree to participate or are disqualified from the study. (If disqualified the oral glucose tolerance test data will be destroyed as well.) This study consists of three parts. The first being phase 1, the second being phase 2, and the third being phase 3. The phase 1 data will stand on its own in the reporting of this study. The long term study is separated into two parts (phase 2 and phase 3) because it is a cross over study, meaning in phase 2 participants will be given either roasted or boiled peanuts (by random assignment) to consume daily for two weeks, then a wash out week will separate phase 2 and 3, and then phase 3 (by the same protocol as phase 2) with the same participants EXCEPT the food treatments will be switched (those who ate roasted peanuts in phase 2 will eat boiled peanuts in phase 3 and vice versa). The data from phase 2 and 3 will be reported together as the experimental design requires each participants to do both treatments. In terms of a time line the phases will be conducted in this order: (Screening and Eligibility - includes 1 oral glucose tolerance test) 1.Phase 1 (includes 2 oral glucose tolerance tests) 2.Wash out week 3.Phase 2 (includes 1 oral glucose tolerance test) 4. Wash out week 5.Phase 3 (includes 1 oral glucose tolerance test) PHASE 1: (2 morning duration in 1 week ~6 hours in lab) Participants will complete an oral glucose tolerance test (OGTT) for the boiled peanut, and roasted peanut treatment (the eligibility oral glucose tolerance test will serve as the control group for phase 1). In the duration of one week the participants will come in on a Wednesday morning for the boiled peanut OGTT and a Friday morning to complete the roasted peanut OGTT. Both OGTT sessions will be conducted as followed: The participants must be fasted when arriving at the lab, meaning they have not eaten in the last 6-8 hours for the scheduled test early in the morning. The participant will consume their treatment food 0 to 15 minutes before consuming the 50g glucose drink. Once the 50 g glucose drink (must be consumed within 10 minuted) is consumed the OGTT will be conducted the same as the eligibility OGTT. The change in blood glucose will be measured over a 2-hr period immediately after consuming the treatment food and 50g glucose drink, blood samples will be taken at 10, 20, 30, 40, 50, 60, 75, 90,120 min using a glucometer to take capillary blood samples (finger-pricks); Investigators will measure height, hip to waist ratio and weight. WASH OUT WEEK: (1 week duration) The participants will return to a free living protocol and will not consume any phase samples (roasted or boiled peanuts) between the phase 1, phase 2 and phase 3. (Participants will be instructed to record all data (exercise/steps and diet) on a paper data collection sheet/diary supplied throughout all phases. At the conclusion of the study during the last glucose tolerance test the participants will hand in their food/exercise diary to Brooke Wilson, the diaries will be immediately transported by her on foot to room 221 of Schaub Hall, locked in a drawer of the graduate office (only Brooke Wilson has the key to the drawer) in which the door to enter the office is locked by a card reader only accessed by associated staff. Investigators will provide a pedometer to participants if they do not have one so they can measure daily activity as a step count. Refer to "19049 information sheet for participant" supporting document for the instructions given to participants on how to use the glucometer, the pedometer, and food restrictions required.) PHASE 2: (2 week duration) Participants will be randomized into the boiled peanut or roasted peanut treatment group. When the participants return to the lab, they will be given the two weeks worth of samples (14 portions of 48 gram servings) for phase 2 (premeasured and separated into individual containers) that they will consume once daily. Depending on the phase, roasted or boiled, they will be instructed on how to properly store the food items to discourage foodborne illness. They will be instructed to consume the sample around the same time everyday between lunch and dinner, to consume in one sitting of 30 minutes instead of throughout the day, and to record the actual time the sample is consumed. PHASE 2 ORAL GLUCOSE TOLERANCE TEST: (1 morning duration ~3 hours in lab) Once the subjects have completed the two weeks of daily x peanut consumption they will complete a oral glucose tolerance test. The participants must be fasted when arrived at the lab, meaning they have not eaten in the last 6-8 hours for the scheduled test early in the morning. The change in blood glucose will be measured over a 2-hr period immediately after consuming a 50g glucose drink. Blood samples will be taken at 10, 20, 30, 40, 50, 60, 75, 90,120 min after consuming the drink using a glucometer to take capillary blood samples (finger-pricks); Investigators will measure height, hip to waist ratio and weight. WASH OUT WEEK: (1 week duration) The participants will return to a completely free living protocol and will not consume any phase samples between phase 2 and phase 3. PHASE 3: (2 week duration) The same procedure for the phase 2 will be used for phase 3 except the groups will switch respective phase samples. PHASE 3 ORAL GLUCOSE TOLERANCE TEST:(1 morning duration ~3 hours in lab) The same procedure for the phase 2 oral glucose tolerance test will be used for phase 3. Investigators will measure height, hip to waist ratio and weight. Throughout the entire procedure the participants may live their life as they normally would except for the following rules. They are strongly discouraged from drinking whatsoever (especially more than 2 drinks per day and or drinking more than 4 drinks in two hours during any time of the study). Also the participants should not do any non habitual exercise less than 10 hours before any oral glucose tolerance test. A phlebotomist is not necessary as the lancing of fingers to obtain enough blood for the glucometer is a common practice and instrument is sold over the counter. As well the glucometer only requires about 50 microliters per finger stick or less, each participant will be required to do five oral glucose tolerance tests including 10 finger lances per test. So in total the greatest amount of blood each participant will draw is 2,500 microliters or the equivalent of 2.5 milliliters. The instruction below of how to properly use a glucose monitor, including lancing of the finger, has been sourced from the Centers for Disease Control and Prevention: -Make sure the glucometer is clean and ready to use, turn on the glucometer. -Wash hands with soap and warm water. Dry well. Massage the hands to get blood into the finger. -Remove the cap off the lancet device, insert lancet until a click is heard to ensure it is secure, twist off the protective top to the lancet exposing the needle and cap the lancet device. -After removing a test strip, immediately close the test strip container tightly. Test strips can be damaged if they are exposed to moisture. -Insert the test strip into the glucometer; check to make sure the glucometer is on. - Place the lancet against the side of the preferred finger; press the button to lance the finger. Prick the finger on the side rather than the tip or pad of finger for less pain. Squeezing from the base of the finger (if it requires a lot of force or no blood is coming out stop and lance again in a different location), gently place a small amount of blood onto the test strip. -After a few seconds, the reading will appear. Track and record the results. -Properly dispose the lancet by removing the lancet device top, recapping the lancet itself and pull the capped lancet out of the device and throw it away. Remove test strip from glucometer and put in appropriate trash container. https://www.cdc.gov/diabetes/managing/managing-blood-sugar/bloodglucosemonitoring.html Pedometer information: PedUSA CW Step Pedometer The pedometer provided only records the amount of steps taken between clearing of data (a button to reset the step count each day). The pedometer does not track any other data than a step count. The participants are allowed to provide their own step counter, in the form of a Fitbit, smart watch, Garmin etc, as long as the device used for the participant is consistent throughout the study. Any step counter apps (not provided) have separate terms of service that may indicate that the users information is shared with third parties that are not the research team, and the information is not confidential. The research team is not responsible for any data shared through these apps as the use of these apps and the awareness and agreement of their terms of use are at the discretion of the participant. *Please refer to the document "MyFitnessPal and Alternative Step Counter Use: Information Related to Personal Data Confidentiality" provided to all participants discussing the data/personal information confidentiality using these technology. * In all situations the participants must physically write down or record their steps in their food diary/exercise diary to be collected by us at the end of each phase. If the pedometer is lost or broken the subject will be provided with a replacement. 50 gram glucose drink information: Azer Scientific Glucose Tolerance Beverages, manufacture # Azer Scientific 10O050, catalog # 22-026-203. The beverage is in compliance with Food and Drug Administration, World Health Organization, and American Diabetes Association. It comes in a premeasured factory sealed bottle ready for consumption and stored at room temperature. Through the course of this study, the participant will spend 15 hours at a lab testing blood glucose levels (in 3-hour sessions) plus 10 minutes per day tracking food and exercise. The total amount of time the participants will spend in this study is 21 hours.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with ages 18 to 65
* BMI ranges [(in kg/m2) 18.5>24.9] from Raleigh-Durham area 3. We will not recruit pregnant women

Exclusion Criteria:

* BMI >24.9 kg/m2 or <18 kg/m2
* Type 1 or 2 diabetes
* Anemia
* Fasting glucose >125 mg/dL
* Use of medication that affect glucose metabolism, renal, liver, pancreatic, or cardiovascular disease.
* Uncontrolled hypertension
* Disorders of the esophageal or in gastrointestinal motility
* Hypo- or hyperthyroidism
* Allergy to peanuts
* Pregnancy.
* Body weight < 110 lb
* Insulin Resistance
* Polycystic Ovary Syndrome
* Food intolerances

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Blood Glucose Response (Glycemic Response) | [week 1 - phase 1 - three measurements mon/wed/fri] [week 2 - wash out week] [week 3 & week 4- phase 2 - one measurement at the end of week 4] [week 5 - wash out week] [week 6 & week 7 - phase 3 - one measurement at end of week 7]
  The blood glucose response will be measured during each oral glucose tolerance test. These tests will happen periodically through out the study to determine if there is any correlation and or significant difference in glycemic response between consuming boiled or roasted peanuts (acute and chronic consumption). The metric is the blood glucose concentration measured by a blood glucose monitor by finger prick 10 times over a two hour period after consuming a standardized 50 gram glucose beverage. The 10 blood glucose measurements are synthesized into one measurement to display a pattern of blood glucose concentrations called the glycemic response.
  Please refer to Study Description -Detailed Description for a more thorough explanation.

SECONDARY OUTCOMES:
weight change | Once week one, once week 4, once week 8.
  Weight of each participant will be measured to determine any weight loss or gain during the study.
waist to hip ratio | Once week one, once week 4, once week 7.
  Waist to hip ration of each participant will be measured to further define any weight change during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Allen, PhD, Study Chair — North Carolina State University; Lisa Dean, PhD, Study Director — USDA ARS - Market Quality and Handling Unit, North Carolina State University
Locations (1):
- North Carolina State University, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The de-identified individual participant data will not be shared unless the study is successful and is published.

DOCUMENTS (1):
  • Informed Consent Form (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT04171648/ICF_000.pdf